CLINICAL TRIAL: NCT05264402
Title: Comparison of Early Phase Infections Risk Between Midline and Piccline Caheters: MIDLINE AND PICCLINE CATHETERS
Acronym: PICCORMID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PICCORMID (29BRC21.0288)
Record Dates: First submitted 2022-01-11; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-01

CONDITIONS: Catheter-related Bloodstream Infection
Keywords: venous access; Midline; PICC line; catheter-related bloodstream infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PICCline group: Patients needing a vascular approach using PICCline catheters
- Midline group: Patients needing a vascular approach using Midline catheters

SUMMARY:
A long-term venous access is frequently required in patient management. Currently, it is ensured by using the long peripheral intravenous catheters (Midline) or peripheral inserted central catheters (PICC line). Either is inserted into a peripheral vein of the upper arm and extends to the distal axillary vein.

If the indications for the two catheters can sometimes be debated, the Midline catheter seems to be more and more used. The complications related to the use of PICC lines have been well described in literature, whereas the comparison of the two catheter-related complications has been less analysed.

The aim of this study is to compare the incidences of catheter-related bloodstream infections linked to PICCs and Midlines.

DETAILED DESCRIPTION:
This single-center observational study will record and compare Midline and PICC line catheter-related bloodstream infections in the first 30 days after placement, catheter-related bloodstream infections being defined as clinical signs associated with a positive catheter culture (bacterial culture finding more than 103 CFU/mL) without any other infectious entry points.

Catheter indications, insertion conditions, incidence of haemorrhagic and thrombotic complications during the first 30 days will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Major ≥ 18 years old
* opposition formulated

Exclusion Criteria:

* Refusal of participation
* Patients under legal protection (guardianship, curatorship, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients requiring a vascular approach using PICCline or Midline catheters
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Compared rate of catheter-related bloodstream infections in the first 30 days in Midline and PICCline group. Catheter-related bloodstream infections are defined as clinical signs with a positive catheter culture without any other infectious entry points. | first 30 days after placement
  catheter-related bloodstream infections being defined as clinical signs (fever, swelling, pain) associated with a positive catheter culture (bacterial culture finding more than 103 CFU/mL) without any other infectious entry points.
  the number of infections recorded will be compared between the group of patients having a Midline and the group of patients having a PICCline

SECONDARY OUTCOMES:
catheter placement time will be evaluated in days | first 30 days after placement
  catheter placement time will be evaluted by measuring the time between catheter placement and removal in days
rate of no infection complications like obstruction, accidental removal, thrombosis, hemorrhagic complications | first 30 days
  The number of mechanical compliaction (obstruction, accidental removal, etc.), haemorrhagic and thrombotic complications recorded will be compared between the group of patients having a Midline and the group of patients having a PICCline

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one year and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.